CLINICAL TRIAL: NCT02859129
Title: An Open-Label, 2-Cohort Study to Evaluate the 2-Way Interaction Between Multiple Doses of Epanova™ and a Single Dose of Rosuvastatin (Crestor®), to Assess the Dose Proportionality of Epanova™, and to Compare the Systemic Exposure of Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) Following Multiple Doses of Epanova™ and Vascepa® in Healthy Normal Subjects
Brief Title: Study to Evaluate the 2-Way Interaction Between Multiple Doses of Epanova™ and a Single Dose of Rosuvastatin (Crestor®)
Acronym: ECLIPSEIII
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OM-EPA-009
Record Dates: First submitted 2016-07-18; First posted 2016-08-08 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Hypertriglyceridemia
Keywords: Epanova; omega-3 carboxylic acids; Vascepa; Eicosapentaenoic acid ethyl ester; Crestor; rosuvastatin
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Rosuvastatin Calcium; Tablets; eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rosuvastatin (Experimental): Single oral dose of 40 mg (1 x 40 mg tablet) rosuvastatin (Crestor®) (Day 1).
  Interventions: Drug: rosuvastatin 40 mg tablet
- Epanova® (Experimental): Multiple oral doses of 2 g (2 x 1 g capsules) Epanova® QD for 10 consecutive days (Days 4 to 13)
  Interventions: Drug: Epanova™ QD (2 x 1 g capsules)
- Epanova® + Crestor® (Experimental): Epanova® multiple oral doses of 4 g (4 x 1 g capsules) QD for 13 consecutive days (Days 14 to 26) with coadministration of single 40 mg (1 x 40 mg tablet) oral dose of rosuvastatin (Crestor®) with the 11th dose of 4 g Epanova® on Day 24
  Interventions: Drug: Multiple doses of 4 g Epanova™ with single of rosuvastatin 40 mg dose
- Vascepa® (Active Comparator): Vascepa® multiple oral doses of 2 g (2 x 1 g capsules) every 12 hours for 20 consecutive days (Days 1 to 20).
  Interventions: Drug: Multiple (20) oral doses of 2 g Vascepa® every 12 hours

INTERVENTIONS:
Drug: rosuvastatin 40 mg tablet — Single oral dose of 40 mg (1 x 40 mg tablet) rosuvastatin (Crestor®) (Day 1).
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Epanova™ QD (2 x 1 g capsules) — Multiple oral doses of 2 g (2 x 1 g capsules) Epanova™ QD for 10 consecutive days (Days 4 to 13)
  Other Names: omega-3 carboxylic acids
  Arms: Epanova®
Drug: Multiple doses of 4 g Epanova™ with single of rosuvastatin 40 mg dose — Multiple oral doses of 4 g Epanova™ QD for 13 consecutive days with coadministration of single 40 mg oral dose of rosuvastatin (Crestor®) with the 11th dose of Epanova™ on Day 24
  Other Names: omega-3 carboxylic acids; Crestor
  Arms: Epanova® + Crestor®
Drug: Multiple (20) oral doses of 2 g Vascepa® every 12 hours — Multiple oral doses of 2 g (2 x 1 g capsules) Vascepa® every 12 hours for 20 consecutive days (Days 1 to 20).
  Other Names: icosapent ethyl
  Arms: Vascepa®

SUMMARY:
This study is intended to evaluate the potential 2-way reciprocal interaction between multiple doses of Epanova™ and a single dose of rosuvastatin

DETAILED DESCRIPTION:
The PK of rosuvastatin will be monitored following single-dose administration of rosuvastatin with and without multiple-dose administration of 4 g Epanova™ for 13 consecutive days in order to detect a possible interaction between rosuvastatin and Epanova™. The PK of total EPA, total DHA and total EPA+DHA will also be monitored following multiple-dose administration of Epanova™ with and without single-dose administration of 40 mg rosuvastatin. A single dose administration for rosuvastatin has been judged sufficient to yield plasma concentrations that will be detectable with an adequate validated analytical method and characterize adequately the PK of rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non-childbearing potential)
* Body Mass Index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at screening
* Non-smoker
* Medically healthy with no clinically significant laboratory profiles, vital signs or ECGs

Exclusion Criteria:

* mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study
* History or presence of myopathy and/or hypothyroidism.
* History or presence of transaminase elevations
* History or presence of hypersensitivity or idiosyncratic reaction to rosuvastatin, to other HMG-CoA reductase inhibitors, to Epanova™, to Vascepa®, or to related compounds
* Known sensitivity or allergy to soybeans, fish, and/or shellfish.
* Has consumed fish within 7 days prior to check-in.
* Female subjects who are pregnant or lactating.
* Positive urine drug and alcohol results at screening or check-in.
* Positive urine cotinine at screening and check-in
* Use of any drugs known to be inducers of CYP enzymes and/or P-gp
* Donation of blood or significant blood loss within 56 days prior to the first dose of study medication.
* Plasma donation within 7 days prior to the first dose of study medication.
* Participation in another clinical trial within 28 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
ln-transformed Cmax,ss of baseline-adjusted total EPA, total DHA, and total EPA+DHA | Days 1 and 24
  ln-transformed Cmax,ss of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA using a linear mixed effect model.
ln-transformed AUC0-tau of baseline-adjusted total EPA, total DHA, and total EPA+DHA | Days 1 and 24
  ln-transformed AUC0-tau of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA using a linear mixed effect model.

SECONDARY OUTCOMES:
ln-transformed Cmax,ss of unadjusted total EPA, total DHA, and total EPA+DHA | Days 1 and 24
  ln-transformed Cmax,ss of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA using a linear mixed effect model.
dose proportionality of baseline-adjusted total EPA, total DHA, and total EPA+DHA systemic exposure will be assessed following multiple doses of Epanova™ 2 g and 4 g | Days 1 and 24
  In Cohort 1 only, dose proportionality of baseline-adjusted total EPA, total DHA, and total EPA+DHA systemic exposure will be assessed following multiple doses of Epanova™ 2 g and 4 g using an analysis of variance (ANOVA) on dose normalized data.
ln-transformed AUC0-tau of unadjusted total EPA, total DHA, and total EPA+DHA | Days 1 and 24
  ln-transformed AUC0-tau of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA using a linear mixed effect model.

OTHER OUTCOMES:
ln-transformed AUC0-24 exposure of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA following multiple doses of Epanova™ compared to multiple doses of Vascepa® | Days 1 and 24
  The systemic exposure of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA following multiple doses of Epanova™ compared to multiple doses of Vascepa® will be assessed by analyzing the ln-transformed AUC0-24. In addition to an ANOVA, an analysis of covariance (ANCOVA) including the baseline value as a covariate will be performed.
AEs, vital signs, ECG, laboratory tests | through study completion (14 days)
  all AEs, physical examinations, vital signs (heart rate, blood pressure, respiratory rate, and temperature), 12-lead ECGs, and laboratory safety tests (hematology, serum chemistry, coagulation, and urinalysis).
ln-transformed Cavg of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA following multiple doses of Epanova™ compared to multiple doses of Vascepa® | Days 1 and 24
  The systemic exposure of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA following multiple doses of Epanova™ compared to multiple doses of Vascepa® will be assessed by analyzing the ln-transformed Cavg. In addition to an ANOVA, an analysis of covariance (ANCOVA) including the baseline value as a covariate will be performed.
ln-transformed Cmax,ss of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA following multiple doses of Epanova™ compared to multiple doses of Vascepa® | Days 1 and 24
  The systemic exposure of baseline-adjusted (primary analysis) and unadjusted (secondary analysis) total EPA, total DHA, and total EPA+DHA following multiple doses of Epanova™ compared to multiple doses of Vascepa® will be assessed by analyzing the ln-transformed Cmax,ss. In addition to an ANOVA, an analysis of covariance (ANCOVA) including the baseline value as a covariate will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Davidson, MD, Study Director — Omthera Pharmaceuticals/AstraZeneca; Sandra M Connolly, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Neptune City, New Jersey, United States

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4425&filename=OMA_EPA_009_CSR.pdf